CLINICAL TRIAL: NCT03433937
Title: Prevention of Seroma Following Inguinal Lymph Node Dissection With Prophylactic Incisional Negative Pressure Wound Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low inclusion
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Mads Gustaf Jørgensen, MD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S-20170085
Record Dates: First submitted 2018-01-30; First posted 2018-02-15 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Seroma; Surgical Site Infection; Lymphedema; Quality of Life
MeSH Terms: conditions — Seroma; Surgical Wound Infection; Lymphedema | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Negative pressure wound therapy (Experimental)
  Interventions: Device: Negative pressure wound therapy
- Control (Active Comparator): Micropore tape
  Interventions: Other: Micropore tape

INTERVENTIONS:
Device: Negative pressure wound therapy — Wound dressing
  Other Names: vacuum assisted closure
  Arms: Negative pressure wound therapy
Other: Micropore tape — Wound dressing
  Arms: Control

SUMMARY:
Inguinal lymph node dissection (ILND) is indicated following metastatic malignant melanoma, and is associated with a high-complication rate, of which many begin with the formation of seroma and ends in complicated wound healing, reoperation, multiple outpatient visits and re-hospitalization. Prevention of seroma may therefore lead to a reduction of many of the preceding complications and improve patient quality-of-life. The aim of this study is to evaluate the efficacy and oncological safety of prophylactic negative pressure wound therapy following ILND in melanoma patients.

ELIGIBILITY:
Inclusion Criteria:

* All malignant melanoma patients who are candidates for ILND and 18 years of age or older

Exclusion Criteria:

* Patients suspected of having tumor residuals after ILND, previous groin irradiation or patients suffering from dementia or any psychiatric disorder making them incapable of informed consent or adherence to follow up, along with patients who are unable to communicate in Danish or English will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with seroma | 3 months
  One or more inguinal seroma(s) which require aspiration

SECONDARY OUTCOMES:
Number of seromas for each participant | 3 months
  Number of aspirated seromas (No.)
Volume of seromas for each participant | 3 months
  Volume of aspirated seromas (mL)
Number of participants with surgical wound infection | 3 months
  Inguinal wound infection which require antibiotic treatment
Number of participants with wound rupture | 3 months
  Inguinal wound rupture which require addition suturing or NPWT treatment
Number of participants with wound necrosis | 3 months
  Inguinal wound necrosis which require debridement
Number of participants with hematoma | 3 months
  Inguinal wound hematoma which require evacuation
Questionnaire EQ-5D-5L | Baseline, 3 months and 2 years
  Quality of life measurement score
Hospitalization time | 3 months
  Length of hospital stay until discharge (days)
Hospitalization readmission time | 3 months
  Length of hospital readmissions (days)
Number of participants with reoperations | 3 months
  Re-operation with opening of the wound or scar under general anesthesia due to adverse complications
Number of participants with lymphedema | 2 years
  Clinical evaluation using the International Lymphedema Society staging
Questionnaire LYMQOL | 2 years
  Lymphedema quality of life measurement score
Number of participants with regional recurrence | 2 years
  Histological verified recurrence to the inguinal site

CONTACTS AND LOCATIONS:
Overall Officials: Jens A Sørensen, Study Chair — Department of Plastic Surgery, Odense University Hospital
Locations (4):
- Denmark (4):
  - Dept. of Plastic Surgery, Rigshospitalet, Copenhagen
  - Dept. of Plastic Surgery, Herlev Gentofte Hospital, Herlev
  - Dept. of Plastic Surgery, Odense University Hospital, Odense
  - Dept. of Plastic Surgery, Roskilde Hospital, Roskilde

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jorgensen MG, Toyserkani NM, Thomsen JB, Sorensen JA. Surgical-site infection following lymph node excision indicates susceptibility for lymphedema: A retrospective cohort study of malignant melanoma patients. J Plast Reconstr Aesthet Surg. 2018 Apr;71(4):590-596. doi: 10.1016/j.bjps.2017.11.026. Epub 2017 Nov 28. PMID 29246739
- [Derived] Jorgensen MG, Chakera AH, Holmich LR, Drejoe JB, Andersen PCL, Khorasani H, Toyserkani NM, Thomsen JB, Sorensen JA. Can prophylactic incisional negative pressure wound therapy Reduce Wound Complications After Inguinal Lymph Node Dissection for Melanoma? Results from a Randomized Controlled Trial. JPRAS Open. 2022 Aug 26;34:134-143. doi: 10.1016/j.jpra.2022.08.003. eCollection 2022 Dec. PMID 36304071
- [Derived] Jorgensen MG, Toyserkani NM, Hyldig N, Chakera AH, Holmich LR, Thomsen JB, Sorensen JA. Prevention of seroma following inguinal lymph node dissection with prophylactic, incisional, negative-pressure wound therapy (SEROMA trial): study protocol for a randomized controlled trial. Trials. 2018 Aug 15;19(1):441. doi: 10.1186/s13063-018-2757-6. PMID 30111378